CLINICAL TRIAL: NCT03757689
Title: Neoadjuvant PD-1 Blockade in Patients with Stage IIB/C Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 09618; 832023 (Other: U Penn IRB); CRU (Other: ACC)
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
Keywords: Stage IIB/C
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; sarcolipin; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Pembrolizumab (Experimental): Subjects will receive one dose of pembrolizumab 200 mg. Approximately 3 weeks after the initial dose of pembrolizumab, subjects will undergo wide excision and sentinel lymph node (SLN) biopsy. Post-operatively, subjects will receive up to 1 year of adjuvant pembrolizumab 200 mg every 3 weeks.
  Interventions: Drug: Pembrolizumab; Procedure: Wide Excision and Sentinel Lymph Node (SLN) Biopsy

INTERVENTIONS:
Drug: Pembrolizumab — Pre-Surgery: Pembrolizumab, one 200mg dose; Post-Surgery: Pembrolizumab, 200 mg every 3 weeks.
Procedure: Wide Excision and Sentinel Lymph Node (SLN) Biopsy — Wide excision and SLN biopsy and pathologic assessment of tissue will be performed per standard of care.

SUMMARY:
The main purpose of this study is to determine the rate of positive sentinel lymph nodes (i.e. the closest draining lymph node(s) to the primary melanoma site) and to test whether treatment with pembrolizumab before surgery to remove melanoma reduces the rate of positive sentinel lymph nodes in patients with Stage IIB/C melanoma.

Subjects with stage II melanoma will receive one dose of pembrolizumab 200 mg, then undergo standard definitive surgery with wide excision and sentinel lymph node (SLN) biopsy approximately 3 weeks after the initial dose of pembrolizumab. Post-operatively, subjects will receive up to 1 year of adjuvant pembrolizumab 200 mg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have clinical stage IIB or IIC resectable MEL. Subjects may not have a diagnosis of uveal or mucosal melanoma.
* Either the subject or the subject's legal representative must be willing and able to provide written informed consent for the trial.
* The subject must be ≥18 years of age on day of signing informed consent.
* The subject must have a performance status of 0 or 1 on the ECOG Performance Scale.
* The subject must demonstrate adequate organ function as defined in Table 1; all screening labs must be performed within 21 days of treatment initiation.
* System Laboratory Value

  * Hematologic

    * ANC ≥1500/mcL
    * Platelets ≥100,000/mcL
    * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
  * Renal

    * Serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR
    * ≥50 mL/min for subject with creatinine levels >1.5 X institutional ULN
  * Hepatic

    * Serum total bilirubin ≤1.5 X ULN OR
    * Direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5 ULN
    * AST (SGOT) and ALT (SPGT) ≤2.5 X ULN OR ≤5 X ULN for subjects with liver metastases
  * Coagulation

    * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female participants:

  * A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
  * Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
  * A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and must be willing to use 2 methods of contraception or abstain from heterosexual intercourse for at least 2 weeks prior to the time of first dose of study medication through 120 days after the last dose of study medication.
  * Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
  * Female subjects of childbearing potential are defined as those women who have not been surgically sterilized or have not been free from menses for >1 year.
* Male participants:

  * Male subjects must agree to follow the contraceptive guidance in Appendix 3 starting with the first dose of study medication, while on study, through 120 days after the last dose of study medication.

Exclusion Criteria:

* Subject has unresectable disease; i.e. in the opinion of the surgical oncologist, all of the subject's melanoma cannot be completely removed with a clear margin.
* A woman of child bearing potential who has a positive urine pregnancy test within 72 hours prior to first dose of study drug (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), interferon, high dose IL-2 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy are an exception to this criterion.
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Subject has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study Day 1.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or requires active treatment. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has evidence of active interstitial lung disease or a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV). (HIV 1/2 antibodies) as determined by medical record review.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection as determined by medical record review.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has severe cardiovascular disease, i.e. arrhythmias, requiring chronic treatment, congestive heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease.
* Has hepatic decompensation (Child-Pugh score >6 [class B and C]).
* Has uncontrolled thyroid dysfunction.
* Has uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
SLN Positivity Rate | 3 Weeks
  To determine the SLN positivity rate and test whether the SLN positivity rate is reduced in high risk stage II patients undergoing neoadjuvant PD-1 blockade.
Safety and Tolerability as measured by observed adverse events. | Approximately 5 Years
  All observed adverse events which occur anytime from the initiation of study therapy to 30 days after the final dose of pembrolizumab will be graded and tabled.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | Approximately 5 Years
  Disease-free survival (DFS) is defined as the time from date of surgery to date of first documented disease progression, death due to any cause or last date that patient was documented to be disease-free (i.e., a scan date).
Overall Survival | Approximately 5 Years
  Overall survival (OS) is defined as the time from date of surgery to date of death due to any cause or last patient contact alive. Both DFS and OS outcomes will be measured from date of surgery to allow us to compare DFS and OS estimates with those of other adjuvant trials.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Karakousis, MD, Principal Investigator — Abramson Cancer Center
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided